CLINICAL TRIAL: NCT03430206
Title: Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) Use in Pediatric Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-43220
Record Dates: First submitted 2018-01-20; First posted 2018-02-12 (Actual); Results first posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Oxygen Deficiency; Desaturation of Blood; Hypoventilation; Anesthesia; Adverse Effect
Keywords: high-flow; nasal cannula; laryngoscopy; otolaryngology; oxygen; desaturation; anesthesia; pediatric
MeSH Terms: conditions — Hypoxia; Hypoventilation

STUDY DESIGN:
Intervention Model Description: Patients are randomized at time of enrollment to either the control or intervention arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (No Intervention): Control subjects will undergo their scheduled procedure and recovery with the usual care. Following recovery from anesthesia, a brief questionnaire will be provided to applicable patients or their parents / guardians / representatives.
- Intervention (Experimental): Treatment subjects will undergo the scheduled procedure, with the difference being that a high-flow nasal cannula will be applied prior to the start of the procedure and removed following the procedure's conclusion. While applied, the cannula will deliver high- flow rate oxygen, air, or a mixture of variable oxygen concentration (21-100%) depending on the surgical conditions and requirements. The rate will be set at 1-2L/kg/min with a maximum of 70L/min. Participants in the treatment arm will then proceed to the recovery area as usual. Following recovery from anesthesia, a brief questionnaire will be provided to applicable patients or their parents / guardians / representatives.
  Interventions: Device: High-flow nasal cannula

INTERVENTIONS:
Device: High-flow nasal cannula — While applied, the cannula will deliver high-flow rate oxygen, air, or a mixture of variable oxygen concentration (21-100%) depending on the surgical conditions and requirements. The rate will be set at 2L/kg/min with a maximum of 70L/min. This will be only for the duration of the surgery or procedure.
  Arms: Intervention

SUMMARY:
THRIVE (Transnasal Humidified Rapid-Insufflation Ventilatory Exchange) refers to the use of high-flow nasal cannula to augment the ability to oxygenate and ventilate a patient under general anesthesia. The use of high-flow nasal cannula oxygen supplementation during anesthesia for surgical procedures has been a recent development in the adult population, with limited data analyzing the pediatric population. This study will determine whether high flow nasal cannula oxygen supplementation during surgical or endoscopic procedures can safely prevent desaturation events in children under anesthesia.

DETAILED DESCRIPTION:
Patients undergoing select procedures in the LPCH operating rooms or ambulatory procedure unit, as identified by review of the daily schedule will be reviewed for potential study enrollment. Study personnel will work with preoperative nurses to identify potential participants. When potential candidates are identified, the investigators will discuss with the surgeon or proceduralist and request that he/she talk with patients about study participation to introduce the idea. On the day of surgery, potential subjects will arrive to preoperative intake areas and proceed through the usual preoperative processes. Once in the preoperative intake area, potential participants will be approached by study personnel at least 30 minutes prior to their scheduled procedure for further explanation of the study and obtaining consent and assent. At this time, potential subjects will be evaluated for interval changes in health that may exclude them from the study. A random number generator will be used to enroll participants into either the usual care (control) or THRIVE (treatment) arm. Control subjects will undergo their scheduled procedure and recovery with the usual care. Treatment subjects will undergo the scheduled procedure, with the difference being that a high-flow nasal cannula will be applied prior to the start of the procedure and removed following the procedure's conclusion. While applied, the cannula will deliver high- flow rate oxygen, air, or a mixture of variable oxygen concentration (21-100%) depending on the surgical conditions and requirements. The rate will be set at 1-2L/kg/min with a maximum of 70L/min. Participants in the treatment arm will then proceed to the recovery area as usual. Following recovery from anesthesia, a brief questionnaire will be provided to applicable patients or their parents/guardians/representatives. The intraoperative vital signs and post-operative course will be analyzed with any patient data stored in a deidentified manner on Stanford- compliant encrypted devices.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients less than or equal to 18 years old undergoing general anesthesia for procedures or surgeries at Lucile Packard Children's Hospital.

Exclusion Criteria:

* Pregnancy, absence of parent or legal guardian able to provide written consent for study participation, anatomical or surgical contraindications (epistaxis, basilar skull fractures or abnormalities, nasal surgery or obstruction, nasal fractures, nasal vascular abnormalities), papillomatosis, tracheostomy, emergent surgery for which application of HFNC might delay surgery or might result in increased aspiration risk.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Caruso, M.D., M.Ed., Principal Investigator — Associate Clinical Professor
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
We are discussing with other facilities conducting research similar in description to or study for a possible multi-center study. If such coordination takes place, we anticipate all deidentified data collected with participating investigators.

REFERENCES:
- [Background] Humphreys S, Rosen D, Housden T, Taylor J, Schibler A. Nasal high-flow oxygen delivery in children with abnormal airways. Paediatr Anaesth. 2017 Jun;27(6):616-620. doi: 10.1111/pan.13151. Epub 2017 Apr 10. PMID 28393433
- [Background] Doyle AJ, Stolady D, Mariyaselvam M, Wijewardena G, Gent E, Blunt M, Young P. Preoxygenation and apneic oxygenation using Transnasal Humidified Rapid-Insufflation Ventilatory Exchange for emergency intubation. J Crit Care. 2016 Dec;36:8-12. doi: 10.1016/j.jcrc.2016.06.011. Epub 2016 Jun 23. PMID 27546740
- [Background] Mir F, Patel A, Iqbal R, Cecconi M, Nouraei SA. A randomised controlled trial comparing transnasal humidified rapid insufflation ventilatory exchange (THRIVE) pre-oxygenation with facemask pre-oxygenation in patients undergoing rapid sequence induction of anaesthesia. Anaesthesia. 2017 Apr;72(4):439-443. doi: 10.1111/anae.13799. Epub 2016 Dec 30. PMID 28035669
- [Background] Humphreys S, Lee-Archer P, Reyne G, Long D, Williams T, Schibler A. Transnasal humidified rapid-insufflation ventilatory exchange (THRIVE) in children: a randomized controlled trial. Br J Anaesth. 2017 Feb;118(2):232-238. doi: 10.1093/bja/aew401. PMID 28100527
- [Background] Gustafsson IM, Lodenius A, Tunelli J, Ullman J, Jonsson Fagerlund M. Apnoeic oxygenation in adults under general anaesthesia using Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) - a physiological study. Br J Anaesth. 2017 Apr 1;118(4):610-617. doi: 10.1093/bja/aex036. PMID 28403407
- [Background] Desai N, Fowler A. Use of Transnasal Humidified Rapid-Insufflation Ventilatory Exchange for Emergent Surgical Tracheostomy: A Case Report. A A Case Rep. 2017 Nov 1;9(9):268-270. doi: 10.1213/XAA.0000000000000589. PMID 28622152

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Control subjects will undergo their scheduled procedure and recovery with the usual standard care.
- THRIVE: Participants received high flow nasal oxygen (THRIVE: active nasal oxygen delivery system).
Period: Overall Study
Arm/Group | Standard of Care | THRIVE
Started | 40 | 38
Completed | 18 | 21
Not Completed | 22 | 17

BASELINE CHARACTERISTICS:
Population: Participants who completed the protocol are included in the analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | THRIVE | Total
Number analyzed (Participants) | 18 | 21 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.1 (4.6) | 6.6 (6.2) | 5.5 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 12 | 13 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 13 | 12 | 25
  Asian | 2 | 3 | 5
  Unknown/Unreported | 3 | 6 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 21 | 39
Percent Oxygen Saturation [Mean (Standard Deviation); unit: Percent Saturation] — Population: 3 participants in the THRIVE group were missing baseline values
  Percent Saturation
    number analyzed (Participants) | 18 | 18 | 36
    (all) | 99.7 (0.6) | 99.3 (1.5) | 99.5 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Surgical Interruptions
Description: Number of surgical interruptions defined by a pause in surgical procedures due to need to intervene, normalized to case length.
Time Frame: Duration of surgery (generally less than 2 hours)
Population: Participants who completed the protocol are included in the analysis
Measure: Mean (95% Confidence Interval); unit: Interruptions
Arm/Group | Standard of Care | THRIVE
Number analyzed (Participants) | 18 | 21
Interruptions | 0.645 [0.308 to 1.35] | 0.302 [0.121 to 0.753]
Statistical Analysis 1: Comparison: Standard of Care vs THRIVE; Test type: Other; p = 0.206, Regression, Negative Binomial

2. Secondary Outcome: Oxygen Desaturation Index
Description: Oxygen desaturation index is defined as the number of times a patient has a 4% decrease in saturation from a 120 second rolling mean for greater than 10 seconds
Time Frame: Duration of surgery (generally less than 2 hours)
Population: Participants who completed the protocol are included in the analysis
Measure: Mean (95% Confidence Interval); unit: Events
Arm/Group | Standard of Care | THRIVE
Number analyzed (Participants) | 18 | 21
Events | 1.09 [0.415 to 2.86] | 0.312 [0.100 to 0.976]
Statistical Analysis 1: Comparison: Standard of Care vs THRIVE; Test type: Other; p = 0.101, Regression, Negative Binomial

3. Secondary Outcome: Number of Oxygen Desaturation Events <90% or Defined by a 5% Fall From Baseline if Baseline Saturation < 94%.
Description: Relative incidence of oxygen desaturation as measured by pulse oximetry by second adjusted for post surgical diagnosis
Time Frame: Duration of surgery (generally less than 2 hours)
Population: Participants who completed the protocol are included in the analysis
Measure: Mean (95% Confidence Interval); unit: Events
Arm/Group | Standard of Care | THRIVE
Number analyzed (Participants) | 18 | 21
Events | 0.536 [0.195 to 1.473] | 0.268 [0.087 to 0.826]
Statistical Analysis 1: Comparison: Standard of Care vs THRIVE; Test type: Other; p = 0.371, Regression, Negative Binomial

4. Secondary Outcome: Incidence of Oxygen Desaturation
Description: Absolute incidence of oxygen desaturation less than 90% as measured by pulse oximetry by second
Time Frame: Duration of surgery (generally less than 2 hours)
Population: This outcome measure was removed from the analysis plan during the course of the study.
Arm/Group | Standard of Care | THRIVE
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Incidence of Adverse Events
Time Frame: Up to 12 hours
Population: Participants who completed the protocol are included in the analysis
Measure: Mean (95% Confidence Interval); unit: Events
Arm/Group | Standard of Care | THRIVE
Number analyzed (Participants) | 18 | 21
Events | 0.183 [0.061 to 0.547] | 0.268 [0.107 to 0.672]
Statistical Analysis 1: Comparison: Standard of Care vs THRIVE; Test type: Other; p = 0.601, Regression, Negative Binomial

6. Secondary Outcome: End-Tidal Carbon Dioxide (ETCO2)
Description: Ventilation was measured with transcutaneous carbon dioxide sensor
Time Frame: Duration of surgery (generally less than 2 hours)
Population: Participants who completed the protocol are included in the analysis
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Standard of Care | THRIVE
Number analyzed (Participants) | 18 | 21
mmHg | 51.6 [46.5 to 56.7] | 52.8 [48.2 to 57.4]
Statistical Analysis 1: Comparison: Standard of Care vs THRIVE; Test type: Other; p = 0.738, Regression, Negative Binomial

7. Other Pre Specified Outcome: Post-surgical Diagnosis
Description: Location of lesion(s) according to post-surgical diagnosis
Time Frame: Duration of surgery (generally less than 2 hours)
Population: Participants who completed the protocol are included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | THRIVE
Number analyzed (Participants) | 18 | 21
Participants
  Supraglottic | 2 | 10
  Infraglottic | 13 | 10
  Both Supraglottic and Infraglottic | 3 | 1

8. Other Pre Specified Outcome: Gas Pain or Bloating
Description: Incidence of gas pain or bloating as measured by post-operative survey
Time Frame: Evaluated postoperatively in post-anesthesia recovery unit prior to discharge, which is about 60 minutes postoperatively.
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Nasal Irritation
Description: Incidence of nasal irritation as measured by post-operative survey
Time Frame: as for outcome 8
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Sinus Pressure / Pain
Description: Incidence of sinus pressure and/or pain as measured by post-operative survey
Time Frame: as for outcome 8
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Headache
Description: Incidence of headache as measured by post-operative survey
Time Frame: as for outcome 8
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Other Adverse Events
Description: Other adverse events as measured by post-operative survey
Time Frame: as for outcome 8
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 12 hours
Arm/Group | Standard of Care | THRIVE
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/38
Other Adverse Events (participants affected / at risk) | 3/40 | 4/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=40) | THRIVE (N=38)
Nausea (Gastrointestinal disorders) | 2 | 2
Sinus Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nose Bleeding (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Emesis (Gastrointestinal disorders) | 1 | 0
Throat Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Unconfirmed

LIMITATIONS AND CAVEATS:
Enrollment did not meet the threshold needed for statistical significance

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/06/NCT03430206/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/06/NCT03430206/SAP_001.pdf